CLINICAL TRIAL: NCT01496092
Title: Effects of Regular Protein Diet Supplemented With Keto Acid on Insulin Resistance In Peritoneal Dialysis Patients
Brief Title: Study of Keto Acid (KA) on Insulin Resistance in Peritoneal Dialysis (PD) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Dong Jie, Institute of Nephrology, Division of Renal, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAPD
Record Dates: First submitted 2011-08-19; First posted 2011-12-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Insulin Resistance
Keywords: Keto Acid; Peritoneal dialysis; Insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Keto Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Keto Acid supplemented with usual protein diet (Experimental)
  Interventions: Drug: Keto Acid
- usual protein diet (No Intervention)

INTERVENTIONS:
Drug: Keto Acid — 12 tablets per day
  Other Names: Compound α-Ketoacid Tablets
  Arms: Keto Acid supplemented with usual protein diet

SUMMARY:
The overarching aim of this proposal is to examine the effects of usual protein diet supplemented with keto acid (KA) on insulin sensitivity in patients on peritoneal dialysis (PD). The investigators will achieve this goal through a randomized controlled trial of administration of usual protein diet plus KA versus usual protein diet alone in patients on peritoneal dialysis (PD) over a period of 6 months. If successful, the results of this study will provide potential avenues for improvement of metabolic profile of patients on PD and possibly improve long-term outcomes such as cardiovascular disease risk and death.

DETAILED DESCRIPTION:
Specific Aims and Significance:

To evaluate the effects of KA plus usual protein diet on basal and stimulated insulin sensitivity in PD patients.

Hypothesis: Administration of KA plus usual protein diet will improve insulin resistance in peritoneal dialysis patients.

To evaluate the influence of KA plus usual protein diet on non-traditional cardiovascular disease (CVD) markers (markers of inflammation and oxidative stress) in PD patients.

Hypothesis: Administration of KA plus usual protein diet will improve markers of inflammation and oxidative stress in PD patients.

Background and Rationale:

Insulin Resistance in Peritoneal Dialysis Patients. Insulin resistance (IR), the reciprocal of insulin sensitivity, describes a state of reduced biological effect for any given concentration of insulin in the plasma. Insulin resistance plays a major pathophysiological role in glucose intolerance and Type 2 diabetes mellitus (T2DM) and is tightly associated with major public health problems including obesity, hypertension, dyslipidemia, and atherosclerotic cardiovascular disease. Insulin resistance, measured by homeostatic model assessment (HOMA-IR), is reported to be common in chronic kidney disease (CKD) patients, including ones on PD and hemodialysis (HD). HOMA-IR is also shown to be an independent predictor of cardiovascular mortality in non-diabetic maintenance HD patients although the pathophysiological link has not been clearly delineated.

A unique aspect of PD that predisposes patients to IR is the inevitable glucose load from the dialysate required for ultrafiltration. Consequently, the prevalence of metabolic syndrome such as hyperglycemia, dyslipidemia and weight gain is increased in PD patients. As an individual component of metabolic syndrome, IR is significantly higher in PD patients than in HD or pre-dialysis patients (47% vs 21% or 26%). Accordingly, improvement of IR could be a potential intervention to decrease the CVD risk and mortality in PD patients. However, only a few investigations have centered on interventions to ameliorate IR in these patients.

Low Protein Diet Supplemented with Keto Acid as a Potential Strategy to Ameliorate Insulin Resistance in PD Patients. Several small scale studies exploring the effects of low protein diet (LPD) plus KA on glucose metabolism indicated that LPD-KA could improve liver and peripheral tissue insulin sensitivity in CKD patients not yet on maintenance dialysis. There are no studies exploring such effects in maintenance dialysis patients, especially in PD patients. One potential mechanism for the improvement in insulin resistance by KA is the reduction of circulating uremic toxins, although the specific elements are not well delineated. In addition, the supplementation of KA might be helpful since plasma total branched-chain amino acid concentrations correlate with glucose tolerance index in dialysis patients. Since the safety of LPD has not been entirely shown in previous studies for PD patients, and our data indicated that DPI < 0.74g/kg/d was harmful in the long-term PD, the investigators will not provide the LPD for improving the IR. However, the exploration of possible benefits of KA plus usual protein intake in PD patients on insulin sensitivity is intriguing.

ELIGIBILITY:
Inclusion Criteria:

* medically stable and receiving stable PD >= 3 months
* age 18-80 years
* body mass index > 18.5
* Kt/v >= 1.7 or Tccr >= 50l/week/1.73m2
* glucose lactate-buffered PD solutions

Exclusion Criteria:

* pregnancy
* intolerance to the study protocols
* severe, unstable, active, or chronic inflammation disease
* chronic use of anti-inflammatory medication
* severe malnutrition
* a high probability of receiving a kidney transplant or transferring to HD within 6 months
* taking anti-inflammatory medication chronically or taking KA during the past one month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | at 0, 12, 24 week after patients start their study prescription
  Insulin sensitivity will be measured using HOMA-IR.

SECONDARY OUTCOMES:
Oxidative stress | at 0, 12, 24 week after patients start their study prescription
  Oxidative stress will be assessed by Plasma OxLDL.
Inflammatory state | at 0, 12, 24 week after patients start their study prescription
  Inflammatory state will be assessed by C-reactive protein, pro-inflammatory cytokine levels (IL-6) and adipokines (leptin and adiponectin).
Endothelial dysfunction | at 0, 12, 24 week after patients start their study prescription
  sICAM and sVCAM will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Jie Dong, Beijing, Beijing Municipality, China